CLINICAL TRIAL: NCT01753375
Title: Role of Vitamin D on the Relapse Rate of Multiple Sclerosis
Brief Title: Role of Vitamin D in Reducing the Relapse Rate in Patients With Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AlJohara M AlQuaiz, M.D. (Other)
Responsible Party: Sponsor-Investigator, AlJohara M AlQuaiz, M.D., Executive Director of "Princess Nora Chair for Women Health Research" , Associate Professor and Consultant Family Physician, Department of Family and Community Medicine, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: E12816
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing rate; Expanded disability status scale; Vitamin D3
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Active Comparator): Administered orally on weekly basis
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): To be administered orally on weekly basis
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 given as 50000 IU orally on weekly basis
  Arms: Vitamin D3
Dietary Supplement: Placebo — Placebo to be given orally on weekly basis
  Arms: Placebo

SUMMARY:
Vitamin D3 supplementation reduces the incidence of multiple sclerosis.Although clinical cross-sectional studies have demonstrated vitamin D3 as a positive mediator in preventing relapses and disease progression, prospective randomized control trials are nevertheless necessary to confirm these statements and to determine the most efficacious, safe, and the minimum required doses. This hypothesis is going to be tested through a randomized triple blinded controlled trial in which after randomization, one group of patients will receive vitamin D and second group will receive placebo. Both groups are going to be followed in a similar way over a period of one year with follow ups at 4, 8 and 12 months. Vitamin D levels is going to be performed at 0,4, 12 month interval. MRI is going to be done at the beginning and end of trial.The number of relapses and the physical disability will be calculated through the Expanded disability status scale (EDSS).

DETAILED DESCRIPTION:
Study Objectives:

* To estimate the prevalence of vitamin D deficiency in Saudi Multiple Sclerosis(MS) patient coming to King Khalid hospital, multiple sclerosis clinic.
* To compare the difference in the relapse rate among Multiple Sclerosis patients who are taking vitamin D3 (50,000 IU per week) versus those who are not taking Vitamin D3 supplements.
* To assess and compare the improvement in the Expanded Disability Status scale and clinical symptoms among those who are taking vitamin D3 versus those who are on placebo

Study Design: A single centre, triple-blinded, parallel randomized placebo controlled trial.

Methods: All eligible patients with clinical definite MS will be assigned a computer-generated Identification number by the statistician and through randomization divided into two groups, one group receiving vitamin D3 (the intervention arm) and other getting placebo (the control arm). All patients will continue with their routine pre-intervention trial treatment for relapse and remission phases of multiple sclerosis. The first treatment group will receive 50,000 IU units of vitamin D3 per week . The control arm patients, instead of vitamin D3 will receive a placebo supplement that looks, smells and tastes the same as the vitamin D3 for 52 weeks. Compliance with the study treatment will be verified by asking the patients about missed doses and by counting used and unused bottles.

All patients will be asked questions related socio-demographic data, vitamin D related dietary products, physical activity questions, exposure to sunlight and variation according to season, use of sunscreen, body coverage when in sunlight and any previous treatment for Multiple Sclerosis, including any vitamin D supplements. Every follow up visit shall include documentation of complete neurologic and medical history and findings. This will be a triple-blinded trial. The patient, the treating physician and the statistician will be masked to the type of treatment each patient receives.Sealed envelopes containing the vitamin D3 or placebo are going to be handed over to the physician with the computer assigned number of the patient. At each follow-up visit all patients will be required to bring their envelopes along with empty/ filled bottles to assess their compliance with the treatment.

The treating physician will follow all the patients at set regular intervals: 0 (baseline), 4, 8, and 12 months to assess the relapses and the EDSS scores and also to check for any adverse effects arising because of the vitamin D3 supplements. Patients who are going to miss their appointment shall be contacted by the project staff to set another appointment in the subsequent week. All patients are going to be emphasized about the importance of these clinical visits and their compliance with the treatment. All patients will be evaluated by the same treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years
* Confirmed Multiple Sclerosis diagnosis according to McDonald criteria
* Stable neurological functioning for at least one month prior to study entry
* Expanded Disability Scale score (EDSS) less than <_4.0
* Must have had one clinical attack in past two years and at least one new silent T2 or gadolinium-enhancing lesion on MRI within the past one year.
* Willing to participate for the entire 52-week period

Exclusion Criteria:

* pregnant or nursing.
* Connective tissue disease (SLE, Sjogren's disease)
* Endocrine disease (hyperthyroidism, hyperparathyroidism)
* Any medical condition predisposing to hypercalcaemia, nephrolithiasis or renal insufficiency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Relapse rate in patients with Multiple Sclerosis | 12 months

SECONDARY OUTCOMES:
Improvement in the expanded disability status scores after receiving vitamin D3 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: AlJohara M AlQuaiz, M.D, Principal Investigator — King Saud University- Medical college
Locations (1):
- Multiple Sclerosis clinic, Department of Neurology, King Khalid Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Cantorna MT, Hayes CE, DeLuca HF. 1,25-Dihydroxyvitamin D3 reversibly blocks the progression of relapsing encephalomyelitis, a model of multiple sclerosis. Proc Natl Acad Sci U S A. 1996 Jul 23;93(15):7861-4. doi: 10.1073/pnas.93.15.7861. PMID 8755567
- [Background] Hayes CE. Vitamin D: a natural inhibitor of multiple sclerosis. Proc Nutr Soc. 2000 Nov;59(4):531-5. doi: 10.1017/s0029665100000768. PMID 11115787
- [Background] Munger KL, Zhang SM, O'Reilly E, Hernan MA, Olek MJ, Willett WC, Ascherio A. Vitamin D intake and incidence of multiple sclerosis. Neurology. 2004 Jan 13;62(1):60-5. doi: 10.1212/01.wnl.0000101723.79681.38. PMID 14718698
- [Background] Kimball SM, Ursell MR, O'Connor P, Vieth R. Safety of vitamin D3 in adults with multiple sclerosis. Am J Clin Nutr. 2007 Sep;86(3):645-51. doi: 10.1093/ajcn/86.3.645. PMID 17823429
- [Background] Shaygannejad V, Janghorbani M, Ashtari F, Dehghan H. Effects of adjunct low-dose vitamin d on relapsing-remitting multiple sclerosis progression: preliminary findings of a randomized placebo-controlled trial. Mult Scler Int. 2012;2012:452541. doi: 10.1155/2012/452541. Epub 2012 Apr 11. PMID 22567287
- [Background] Jagannath VA, Fedorowicz Z, Asokan GV, Robak EW, Whamond L. Vitamin D for the management of multiple sclerosis. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD008422. doi: 10.1002/14651858.CD008422.pub2. PMID 21154396
- [Background] Burton JM, Kimball S, Vieth R, Bar-Or A, Dosch HM, Cheung R, Gagne D, D'Souza C, Ursell M, O'Connor P. A phase I/II dose-escalation trial of vitamin D3 and calcium in multiple sclerosis. Neurology. 2010 Jun 8;74(23):1852-9. doi: 10.1212/WNL.0b013e3181e1cec2. Epub 2010 Apr 28. PMID 20427749